CLINICAL TRIAL: NCT04930055
Title: Immune Responses in Oncology Patients to Novel Coronavirus Vaccines (IROC)
Status: Terminated | Type: Observational
Why Stopped: PI had decided to terminate the study
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Utpal P. Davé, Associate Professor Department of Medicine Division of Hematology/Oncology, Indiana University
Other Study IDs: CTO-IUSCCC-0759
Record Dates: First submitted 2021-06-15; First posted 2021-06-18 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Cancer
Keywords: COVID-19; Vaccine; Pfizer; Moderna; Janssen; COVID
MeSH Terms: conditions — Neoplasms; COVID-19 | interventions — heterologous prime boost COVID-19 vaccination; 2019-nCoV Vaccine mRNA-1273; Ad26COVS1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Collection at Dose 1, Dose 2, and +1 month, +3 months, +6 months and +12 months after their Dose 2 and/or at booster dose and +1 month, +3 months, +6 months and +12 months after their booster dose for Pfizer/Moderna vaccinations. Collection at Dose 1 and +1 month, +3 months, +6 months and +12 months after their Dose 1 and/or at booster dose and +1 month, +3 months, +6 months and +12 months after their booster dose for Janssen vaccinations.
  PBMC Collection at Dose 1 and +3 months after Dose 2 for Moderna/Pfizer vaccinations and at Dose 1 and +3 months after Dose 1 for Janssen vaccinations and/or at booster dose and +6 months after booster dose of either.
  Serum and peripheral blood mononuclear cells (PBMC) will be cryopreserved for molecular and immunologic studies that can include, but are not limited, to antibody titers, cytokines and chemokines, immune cell subsets and T cell and B cell analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Group 1: Patients with solid tumors receiving courses of cytotoxic therapy.
  Interventions: Biological: COVID-19 Vaccination
- Group 2: Patients with hematological cancers receiving courses of cytotoxic chemotherapy.
  Interventions: Biological: COVID-19 Vaccination
- Group 3: Patients with solid tumors receiving TKIs or other targeted therapies, but not cytotoxic regimens within 3 months
  Interventions: Biological: COVID-19 Vaccination
- Group 4: Patients with hematologic cancers receiving TKIs or other targeted therapies, but not cytotoxic regimens within 3 months
  Interventions: Biological: COVID-19 Vaccination
- Group 5: Patients receiving immune checkpoint inhibitors.
  Interventions: Biological: COVID-19 Vaccination
- Group 6: Patients who underwent allogeneic stem cell transplant within 12 months.
  Interventions: Biological: COVID-19 Vaccination
- Group 7: Patients who underwent cellular therapy, including CAR-T cells or T cells with engineered TCRs within 12 months.
  Interventions: Biological: COVID-19 Vaccination
- Group 8: Patients in remission who have received cellular therapy more than 12 months in the past, including allogeneic, autologous or engineered cellular approaches
  Interventions: Biological: COVID-19 Vaccination
- Group 9: Patients with cancer in remission for at least 2 years not receiving active cytotoxic cancer chemotherapy (hormonal therapy is permitted).
  Interventions: Biological: COVID-19 Vaccination
- Group 10: Patients who have undergone allogenic bone marrow transplant and are currently receiving immunosuppressants
  Interventions: Biological: COVID-19 Vaccination
- Group 11: Patients who have undergone allogenic bone marrow transplant who are not currently receiving immunosuppressants
  Interventions: Biological: COVID-19 Vaccination
- Group 12: Patients who have a cancer diagnosis but do not fall into group 1-11
  Interventions: Biological: COVID-19 Vaccination

INTERVENTIONS:
Biological: COVID-19 Vaccination — Subjects will receive either the Moderna (mRNA-1273), Pfizer (BTN162b2), or Janssen (Ad26.COV2.S) vaccination per standard of care
  Other Names: Moderna (mRNA-1273); Pfizer (BTN162b2); Janssen (Ad26.COV2.S)

SUMMARY:
The goals of this study are to assess initial or booster vaccine performance (safety and efficacy) and to collect serum and peripheral blood mononuclear cells (PBMCs) pre and post-vaccination to assess immune and other response parameters following immunization in cancer patients receiving either the Pfizer (BTN162b2), Moderna (mRNA-1273), or the Janssen (Ad26.COV2.S) vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent and HIPAA authorization
2. Patients deemed eligible and willing to receive a COVID-19 vaccine by treating physician per standard of care.
3. Subjects must be ≥ 18 years old at the time of consent.
4. Diagnosis of cancer and fall into one of the groups below:

   1. Group 1: Patients with solid tumors receiving courses of cytotoxic therapy.
   2. Group 2: Patients with hematological cancers receiving courses of cytotoxic chemotherapy.
   3. Group 3: Patients with solid tumors receiving tyrosine kinase inhibitors (TKIs) or other targeted therapies, but not cytotoxic regimens within 3 months.
   4. Group 4: Patients with hematologic cancers receiving TKIs or other targeted therapies, but not cytotoxic regimens within 3 months.
   5. Group 5: Patients receiving immune checkpoint inhibitors.
   6. Group 6: Patients who underwent allogeneic stem cell transplant within 12 months.
   7. Group 7: Patients who underwent cellular therapy, including Chimeric antigen receptor t-cells (CAR-T) cells or t-cells with engineered t-cell receptors (TCRs) within 12 months.
   8. Group 8: Patients in remission who have received cellular therapy more than 12 months in the past, including allogeneic, autologous or engineered cellular approaches.
   9. Group 9: Patients with cancer in remission for at least 2 years not receiving active cytotoxic cancer chemotherapy (hormonal therapy is permitted).
   10. Group 10: Patients who have undergone allogenic bone marrow transplant and are currently receiving immunosuppressants
   11. Group 11: Patients who have undergone allogenic bone marrow transplant who are not currently receiving immunosuppressants
   12. Group 12: Patients who have a cancer diagnosis but do not fall into group 1-11

3. Estimated survival of 8 weeks or more following enrollment on the study.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active COVID-19 infection or influenza-like-illness. If subjects have previously tested positive for COVID-19 infection, they are eligible to participate in this study after 90 days
2. Unwilling or unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a current or previous cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 2206 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Adverse Event Collection | from date of vaccination until 2 months after full vaccination

SECONDARY OUTCOMES:
Incidence of COVID-19 infection | from date of vaccination until 6 months after full vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Utpal Dave, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Health Joe and Shelly Schwarz Cancer Center, Carmel, Indiana
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No